CLINICAL TRIAL: NCT01191905
Title: Effects of HIgh Volume COntinuous REnal Replacement Therapy in Patients With Septic Acute Kidney Injury
Acronym: HICORES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Gambro Renal Products, Inc. (Industry)
Responsible Party: Principal Investigator, Dong Ki Kim, M.D, PhD, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSGAM-001
Record Dates: First submitted 2010-08-29; First posted 2010-08-31 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Sepsis; Kidney Failure, Acute; Renal Replacement Therapy
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose CRRT (Experimental): Clearance of 80 mL/Kg/hr (1:1 balanced pre-dilution CVVHDF)
  Interventions: Drug: high dose CRRT
- Conventional dose CRRT (Active Comparator): clearance of 40 mL/Kg/hr (1:1 balanced pre-dilution CVVHDF)
  Interventions: Drug: Conventional dose CRRT

INTERVENTIONS:
Drug: high dose CRRT — clearance of 80 mL/Kg/hr (1:1 balanced pre-dilution CVVHDF)
  Arms: High dose CRRT
Drug: Conventional dose CRRT — clearance of 40 mL/Kg/hr (1:1 balanced pre-dilution CVVHDF)
  Arms: Conventional dose CRRT

SUMMARY:
Acute kidney injury (AKI) is a common and serious problem in critically ill patients, and is known to be an independent risk factor for mortality. Among the various etiologies of AKI, sepsis or septic shock is the most frequent contributing factor especially in an intensive care unit setting. Also, the mortality of septic AKI in these patients still remains extremely high despite recent marked therapeutic advance.

Given the physiologic superiority of continuous renal replacement therapy (CRRT) on uremia and volume control, it has become the modality of choice in critically ill patients with AKI. In addition, CRRT can theoretically provide immunohomeostasis through the convective and adsorptive removal of various immune mediators. Although the pathophysiology of septic AKI remains elusive, it has become increasingly recognized that many pro- and anti-inflammatory mediators, such as TNF, IL-6, IL-8 and IL-10, play an important role in this process. Therefore, it has been speculated that the reduction of cytokines by increasing CRRT dose in patients with septic AKI may reduce mortality risk. Even though recent two large scale randomized controlled trials, ATN and RENAL study, have failed to show the difference in survival rate between the clearance of 20~25 ml/kg/hr and 35~40 ml/kg/hr, none of these studies were designed to elucidate the survival benefit of high intensity CRRT in patients with septic AKI. Moreover, the optimal target CRRT dose in these patients is not well established and may be even higher than 35~40 ml/kg/hr in terms of septic AKI. Indeed, recent several uncontrolled trial have shown the survival benefit of high intensity CRRT in these patients.

To further explore the effects of high dose CRRT on survival of critically ill patients with septic AKI, the investigators will conduct a multicenter prospective randomized controlled open-label trial which compares the difference in survival rate between 1:1 balanced pre-dilution CVVHDF at 80 vs. 40 mL/Kg/hr for initial 72hrs after the start of CRRT. The primary end-point of this study is the effect of high volume pre-dilution CVVHDF on 28-day survival rate. The secondary end-point is 60- and 90-day mortality, ICU and in-hospital mortality, duration of CRRT and renal replacement therapy, duration of mechanical ventilation, cytokine removal rate at 12h after the initiation of CRRT, and changes in SOFA and APACHE II score at 72h after the initiation of CRRT. This is a superiority trial which aims to demonstrate a reduction of 20% or more in mortality rate. For this purpose, at least 109 subjects (a total of 218) would be required for each group if type I error rate is 5% and type II error is 20% given 25% of drop-out rate during the study period. Block randomization will be used by means of a dedicated website.

There are still conflicting data on the optimal target dose of CRRT in patients with septic AKI. Our study will address this issue to answer the unresolved question on the effect of high dose CRRT.

ELIGIBILITY:
Inclusion Criteria:

* Consensus criteria for sepsis
* Injury stage of RIFLE criteria or more (>2-fold increase in the serum creatinine or urine output <0.5 mL/kg/hr for 12 hours)
* Absence of other established non-sepsis-related cause of AKI
* written informed consent

Exclusion Criteria:

* patient age < 20 years or > 80 years
* life expectancy less than 3 months (ex. terminal stage of malignancy)
* Child-Pugh class C liver cirrhosis
* Pregnancy or lactation
* History of dialysis prior to the randomization

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Overall mortality | 0 to 28 days

SECONDARY OUTCOMES:
60-day mortality | 0 to 60 days
90-day mortality | 0 to 90 days
ICU mortality | 0 to 90 days
In-hospital mortality | 0 to 90 days
duration of CRRT | 0 to 90 days
duration of renal replacement therapy | 0 to 90 days
duration of mechanical ventilation | 0 to 90 days
cytokine removal rate | 0 to 12h
changes in SOFA and APACHE II score | 0 to 72 hr
hemofilter circuit life | 0 to 72 hr]

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Hyun Yoo, MD, PhD, Study Chair — Yonsei University; Dong Ki Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (5):
- South Korea (5):
  - National Health Insurance Corporation Ilsan Hospital, Koyang
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Seoul National University Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Fayad AI, Buamscha DG, Ciapponi A. Timing of kidney replacement therapy initiation for acute kidney injury. Cochrane Database Syst Rev. 2022 Nov 23;11(11):CD010612. doi: 10.1002/14651858.CD010612.pub3. PMID 36416787
- [Derived] Tsujimoto Y, Miki S, Shimada H, Tsujimoto H, Yasuda H, Kataoka Y, Fujii T. Non-pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2021 Sep 14;9(9):CD013330. doi: 10.1002/14651858.CD013330.pub2. PMID 34519356